CLINICAL TRIAL: NCT02821702
Title: Fertility Post Preservative Cesarean Section and Uterine Artery Embolization
Brief Title: Fertility Post Placenta Accrete
Acronym: CSAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Aya Mohr-Sasson, Doctor, Sheba Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 3178-16- SMC
Record Dates: First submitted 2016-06-17; First posted 2016-07-01 (Estimated); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Fertility
Keywords: placenta accreta; cesarean section; artery embolization
MeSH Terms: conditions — Placenta Accreta | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Post surgery and embolization (Experimental): Blood sample for hormonal profile: estrogen , progesterone, anti mullarian hormone ( AMH) Vaginal ultrasound to estimate antral follicle count ( AFC)
  Interventions: Device: Vaginal ultrasound; Biological: Blood sample
- Control group (Active Comparator): Blood sample for hormonal profile: estrogen , progesterone, anti mullarian hormone ( AMH) Vaginal ultrasound to estimate antral follicle count ( AFC)
  Interventions: Device: Vaginal ultrasound; Biological: Blood sample
- Post surgery with accreta without embolization (Active Comparator): Blood sample for hormonal profile: estrogen , progesterone, anti mullarian hormone ( AMH) Vaginal ultrasound to estimate antral follicle count ( AFC)
  Interventions: Device: Vaginal ultrasound; Biological: Blood sample
- Post surgery without accreta without embolization (Active Comparator): Blood sample for hormonal profile: estrogen , progesterone, anti mullarian hormone ( AMH)
  Interventions: Biological: Blood sample
- Normal Vaginal Delivery - no suspected accreta (Active Comparator): Blood sample for hormonal profile: estrogen , progesterone, anti mullarian hormone ( AMH)
  Interventions: Biological: Blood sample

INTERVENTIONS:
Device: Vaginal ultrasound
  Arms: Control group; Post surgery and embolization; Post surgery with accreta without embolization
Biological: Blood sample

SUMMARY:
This study is the first to investigate the fertility outcome and the influence on ovarian reserve after using uterine artery embolization during cesarean delivery.

DETAILED DESCRIPTION:
Placenta accreta is an abnormal adherence of the placenta to the uterine wall. Three variants of abnormally invasive placentation have been described: placenta accreta, in which placental villi invade the surface of the myometrium; placenta increta, in which placental villi extend into the myometrium; and placenta percreta, where the villi penetrate through the myometrium to the uterine serosa and may invade adjacent organs, such as the bladder.

Placenta accrete is an increasingly prevalent and potentially dangerous complication of pregnancy. It appears to be most strongly predicted by a history of cesarean deliveries and low-lying placenta/previa. Additional risk factors include in vitro fertilization pregnancy, prior myomectomy, Asherman's syndrome, submucous leiomyomata, maternal age older than 35 years, elevated second-trimester levels of α-fetoprotein and β-human chorionic gonadotropin.

Pregnancies complicated with placenta accrete are associated with adverse maternal outcomes, including life-threatening maternal haemorrhage, large-volume blood transfusion, uterine rupture and peripartum hysterectomy. Moreover , strong association was found between abnormal placentation to significant perinatal morbidity and mortality such as small for gestational age, preterm delivery, neonatal intensive care unit hospitalization, perinatal death and neonatal death.

Prenatal diagnosis and adequate planning, particularly in high-risk populations, is indicated for the reduction of these adverse outcomes. Advances in grayscale and Doppler ultrasound have facilitated prenatal diagnosis. Despite advances in imaging techniques, no diagnostic technique affords the clinician complete assurance of the presence or absence of placenta accreta.

Management of placenta accrete could be conservative (aiming for uterine preservation) or interventional ( elective cesarean hysterectomy ) depending on the patients will to maintain the uterus for future fertility, the degree of placentation abnormality or complications during delivery. The extent (area, depth) of the abnormal attachment will determine the response-curettage, wedge resection, medical management, or hysterectomy. Uterine conserving options may work in small focal accretas, but abdominal hysterectomy usually is the most definitive treatment.

Post-partum hemorrhage is the major concern dealing with placenta accrete. Women with placenta accreta have a higher incidence of postpartum hemorrhage and are more likely to undergo emergency hysterectomy .

If the diagnosis or a strong suspicion is formed before delivery, a number of measures should be taken including counseling the patient about the likelihood of hysterectomy and blood transfusion, preparing blood products and clotting factors and considering using cell saver technology.The appropriate location and timing for delivery should be considered to allow access to adequate surgical personnel and equipment and a preoperative anesthesia assessment should be obtained.

A patient with stable vital signs and persistent bleeding, especially if the rate of loss is not excessive, may be a candidate for arterial embolization. Radiographic identification of bleeding vessels allows embolization with gelfoam, coils, or glue. Balloon occlusion is also a technique used in such circumstances. Embolization can be used for bleeding that continues after hysterectomy or can be used as an alternative to hysterectomy to preserve fertility.

Studies estimating the fertility and pregnancy outcomes after successful conservative treatment for placenta accrete have demonstrated placenta accreta does not appear to compromise the patients' subsequent fertility or obstetrical outcome.

By reviewing the literature, no prospective studies have specifically evaluated fertility, following uterine artery embolization during cesarean section due to placenta accrete .

Methods:

Women that were operated and fit inclusion criteria will be invited to participate in the study after getting advanced notice on requirements . After giving informed consent to participate in the study, demographic parameters and medical history will be taken, including - age , Body Mass Index ( BMI), parity, gravity, past medical history, past operations.

preoperative intra operative and post operative information will be collected.

All women participating will complete -

1. Day 2 blood sample for hormonal profile - follicle stimulating hormone ( FSH), estrogen (E2), progesterone (P)
2. Blood sample for anti mullarian hormon (AMH)
3. Vaginal ultrasound assessing antral follicle count (AFC)

ELIGIBILITY:
Inclusion Criteria:

Study group

* S/P cesarean section with bilateral uterine arteries embolization.
* Age 18-42

Control group ( from IVF clinic)

* infertility treatment due to male factor
* Single patients for sperm donation
* Age 18-42

Exclusion Criteria:

* Age >42
* Hysterectomy due to the procedure

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 135 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Ovarian reserve estimated by laboratory test ( Blood sample for AMH) | Through study completion - estimated time is six month
Ovarian reserve estimated by ultrasound evaluation (AFC) | Through study completion - estimated time is six month

CONTACTS AND LOCATIONS:
Overall Officials: Aya Mohr Sasson, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fitzpatrick KE, Sellers S, Spark P, Kurinczuk JJ, Brocklehurst P, Knight M. The management and outcomes of placenta accreta, increta, and percreta in the UK: a population-based descriptive study. BJOG. 2014 Jan;121(1):62-70; discussion 70-1. doi: 10.1111/1471-0528.12405. Epub 2013 Aug 7. PMID 23924326
- [Background] Eshkoli T, Weintraub AY, Sergienko R, Sheiner E. Placenta accreta: risk factors, perinatal outcomes, and consequences for subsequent births. Am J Obstet Gynecol. 2013 Mar;208(3):219.e1-7. doi: 10.1016/j.ajog.2012.12.037. Epub 2013 Jan 8. PMID 23313722
- [Background] Balayla J, Bondarenko HD. Placenta accreta and the risk of adverse maternal and neonatal outcomes. J Perinat Med. 2013 Mar;41(2):141-9. doi: 10.1515/jpm-2012-0219. PMID 23241664
- [Background] Clark SL, Koonings PP, Phelan JP. Placenta previa/accreta and prior cesarean section. Obstet Gynecol. 1985 Jul;66(1):89-92. PMID 4011075
- [Background] Oyelese Y, Smulian JC. Placenta previa, placenta accreta, and vasa previa. Obstet Gynecol. 2006 Apr;107(4):927-41. doi: 10.1097/01.AOG.0000207559.15715.98. PMID 16582134
- [Background] Vahanian SA, Lavery JA, Ananth CV, Vintzileos A. Placental implantation abnormalities and risk of preterm delivery: a systematic review and metaanalysis. Am J Obstet Gynecol. 2015 Oct;213(4 Suppl):S78-90. doi: 10.1016/j.ajog.2015.05.058. PMID 26428506
- [Background] Rao KP, Belogolovkin V, Yankowitz J, Spinnato JA 2nd. Abnormal placentation: evidence-based diagnosis and management of placenta previa, placenta accreta, and vasa previa. Obstet Gynecol Surv. 2012 Aug;67(8):503-19. doi: 10.1097/OGX.0b013e3182685870. PMID 22926275
- [Background] Zaki ZM, Bahar AM, Ali ME, Albar HA, Gerais MA. Risk factors and morbidity in patients with placenta previa accreta compared to placenta previa non-accreta. Acta Obstet Gynecol Scand. 1998 Apr;77(4):391-4. PMID 9598946
- [Derived] Mohr-Sasson A, Haas J, Bar-Adon S, Shats M, Hochman R, Orvieto R, Mazaki-Tovi S, Sivan E. The Influence of Cesarean Delivery on Ovarian Reserve: a Prospective Cohort Study. Reprod Sci. 2022 Feb;29(2):639-645. doi: 10.1007/s43032-021-00730-z. Epub 2021 Sep 1. PMID 34472035